CLINICAL TRIAL: NCT06121323
Title: Physiological Effects of Lactate in Individuals With Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henrik Wiggers (Other)
Responsible Party: Sponsor-Investigator, Henrik Wiggers, Professor, Senior Consultant, MD, PhD, DMSc, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: LACTATE-CHF
Record Dates: First submitted 2023-09-20; First posted 2023-11-07 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure, Systolic
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactate infusion (Active Comparator): All participants will be randomized to first receive a three-hour intravenous infusion with either a racemic (D/L) mixture of sodium lactate or intravenous isotonic sodium chloride placebo. All participants will then cross over to the converse infusion on the same day.
  Interventions: Other: Sodium lactate infusion
- Lactate ingestion (Active Comparator): All participants will be randomized to first receive either an orally administered racemic (D/L) mixture of sodium lactate or isocaloric, isovolumic oral placebo (maltodextrin). The oral dose of lactate will be equal to the intravenous dose. All participants will be studied for three hours and then cross over to receive the converse oral administration following additional three hours of observation time on the same day.
  Interventions: Other: Sodium lactate ingestion

INTERVENTIONS:
Other: Sodium lactate infusion — Dosage of sodium-lactate: 0.5 mol/L; 3 mL/kg/time; maximal 300 mL/hour.
  Arms: Lactate infusion
Other: Sodium lactate ingestion — Oral dose is equal to the i.v. dose.
  Arms: Lactate ingestion

SUMMARY:
Background:

Lactate is continuously produced in the human body through two primary processes: glycolysis and microbial fermentation in the gastrointestinal tract. At rest, its concentration in the bloodstream typically ranges from 1 to 2 mmol/L. However, during periods of physical exertion or insufficient oxygen supply, such as during intense exercise, lactate levels significantly increase. Traditionally, lactate was perceived as a byproduct of anaerobic metabolism. Nevertheless, emerging research has illuminated its vital role as both a signaling molecule and a crucial energy source for vital organs like skeletal muscle, brain, and the heart.

Objectives:

The primary aim of this study is to investigate the impact of physiological levels of circulating lactate on the hemodynamics of individuals with chronic heart failure. This research seeks to understand how lactate affects the cardiovascular response in this specific patient population.

Design and Endpoints:

The study design employs a double-blind, randomized crossover approach involving 12 heart failure patients. Each participant will undergo two separate visits.

Visit 1: Participants will receive a three-hour intravenous infusion of either a racemic (D/L) mixture of sodium lactate or an intravenous isotonic sodium chloride placebo, with a subsequent crossover to the opposite infusion on the same day.

Visit 2: Similar to the first visit, participants will receive either an orally administered racemic (D/L) mixture of sodium lactate or an isocaloric, isovolumic oral placebo (maltodextrin), with a crossover to the opposite administration after three hours.

The study's endpoints include cardiac output (primary), mixed venous saturation (SVO2), pulmonary wedge pressure, resting echocardiography (left ventricular ejection fraction and myocardial work efficiency), and measurements of vasoactive substances in blood samples.

Methods:

The study employs invasive Swan-Ganz monitoring to measure cardiac output, echocardiography, and frequent venous blood sample collections. These measurements and samples will be taken at specific intervals during the study visits.

Intervention:

To investigate the isolated hemodynamic and physiological effects of lactate, the study utilizes lactate infusion and ingestion to induce a state of hyperlactatemia within the physiological range. The intended dosages aim to stay within the physiological range, with no values expected to exceed 3-4 mmol/L.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure
* NYHA II-III
* Left ventricular ejection fraction <40%
* Negative urine-HCG for women with childbearing potential

Exclusion Criteria:

* Diabetes or HbA1c >48 mmol/mol
* Significant cardiac valve disease
* Severe stable angina pectoris
* Severe comorbidity as judged by the investigator
* Inability to give informed consent
* Age <18 years
* Other disease or treatment making subject unsuitable for study participation as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2025-01-16 (Actual)

PRIMARY OUTCOMES:
Cardiac output Cardiac output | Two visits of six hours each separated by a one-week washout period. Thus, outcome measures for the intravenous route will be assessed at week one, and outcome measures for the oral route will be assessed at week 2.
  Unit: L/min.
  It represents the amount of blood that the heart pumps out of the left ventricle per minute.

SECONDARY OUTCOMES:
Mixed venous saturation (SVO2) | Two visits of six hours each separated by a one-week washout period. Thus, outcome measures for the intravenous route will be assessed at week one, and outcome measures for the oral route will be assessed at week 2.
  Unit: %
  It represents the percentage of oxygen saturation in the blood as it returns to the right side of the heart after circulating through the body's tissues.
Pulmonary wedge pressure | Two visits of six hours each separated by a one-week washout period. Thus, outcome measures for the intravenous route will be assessed at week one, and outcome measures for the oral route will be assessed at week 2.
  Unit: mmHg
  It reflects the pressure within the left atrium and the left ventricle of the heart, and it is an important indicator of left ventricular preload.
Left ventricular ejection fraction | Two visits of six hours each separated by a one-week washout period. Thus, outcome measures for the intravenous route will be assessed at week one, and outcome measures for the oral route will be assessed at week 2.
  Unit: %
  It is a measure of the percentage of blood that is pumped out of the left ventricle with each heartbeat.
Global longitudinal strain | Two visits of six hours each separated by a one-week washout period. Thus, outcome measures for the intravenous route will be assessed at week one, and outcome measures for the oral route will be assessed at week 2.
  Unit: %
  It quantifies the deformation or shortening of the heart muscle fibers along the longitudinal (lengthwise) axis of the left ventricle during the cardiac cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Wiggers, Professor, Study Chair — Dept. of Cardiology, Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goodwin ML, Harris JE, Hernandez A, Gladden LB. Blood lactate measurements and analysis during exercise: a guide for clinicians. J Diabetes Sci Technol. 2007 Jul;1(4):558-69. doi: 10.1177/193229680700100414. PMID 19885119
- [Background] Vincent JL, Quintairos E Silva A, Couto L Jr, Taccone FS. The value of blood lactate kinetics in critically ill patients: a systematic review. Crit Care. 2016 Aug 13;20(1):257. doi: 10.1186/s13054-016-1403-5. PMID 27520452
- [Background] Brooks GA. The tortuous path of lactate shuttle discovery: From cinders and boards to the lab and ICU. J Sport Health Sci. 2020 Sep;9(5):446-460. doi: 10.1016/j.jshs.2020.02.006. Epub 2020 Feb 21. PMID 32444344
- [Background] Johannsson E, Lunde PK, Heddle C, Sjaastad I, Thomas MJ, Bergersen L, Halestrap AP, Blackstad TW, Ottersen OP, Sejersted OM. Upregulation of the cardiac monocarboxylate transporter MCT1 in a rat model of congestive heart failure. Circulation. 2001 Aug 7;104(6):729-34. doi: 10.1161/hc3201.092286. PMID 11489783
- [Background] Liu C, Wu J, Zhu J, Kuei C, Yu J, Shelton J, Sutton SW, Li X, Yun SJ, Mirzadegan T, Mazur C, Kamme F, Lovenberg TW. Lactate inhibits lipolysis in fat cells through activation of an orphan G-protein-coupled receptor, GPR81. J Biol Chem. 2009 Jan 30;284(5):2811-2822. doi: 10.1074/jbc.M806409200. Epub 2008 Dec 1. PMID 19047060
- [Background] Offermanns S. Hydroxy-Carboxylic Acid Receptor Actions in Metabolism. Trends Endocrinol Metab. 2017 Mar;28(3):227-236. doi: 10.1016/j.tem.2016.11.007. Epub 2017 Jan 10. PMID 28087125
- [Background] Engelstoft MS, Park WM, Sakata I, Kristensen LV, Husted AS, Osborne-Lawrence S, Piper PK, Walker AK, Pedersen MH, Nohr MK, Pan J, Sinz CJ, Carrington PE, Akiyama TE, Jones RM, Tang C, Ahmed K, Offermanns S, Egerod KL, Zigman JM, Schwartz TW. Seven transmembrane G protein-coupled receptor repertoire of gastric ghrelin cells. Mol Metab. 2013 Sep 4;2(4):376-92. doi: 10.1016/j.molmet.2013.08.006. eCollection 2013. PMID 24327954
- [Background] Pedersen MGB, Sondergaard E, Nielsen CB, Johannsen M, Gormsen LC, Moller N, Jessen N, Rittig N. Oral lactate slows gastric emptying and suppresses appetite in young males. Clin Nutr. 2022 Feb;41(2):517-525. doi: 10.1016/j.clnu.2021.12.032. Epub 2021 Dec 24. PMID 35016146
- [Background] Nalos M, Leverve X, Huang S, Weisbrodt L, Parkin R, Seppelt I, Ting I, Mclean A. Half-molar sodium lactate infusion improves cardiac performance in acute heart failure: a pilot randomised controlled clinical trial. Crit Care. 2014 Mar 25;18(2):R48. doi: 10.1186/cc13793. PMID 24666826
- [Background] Leverve XM, Boon C, Hakim T, Anwar M, Siregar E, Mustafa I. Half-molar sodium-lactate solution has a beneficial effect in patients after coronary artery bypass grafting. Intensive Care Med. 2008 Oct;34(10):1796-803. doi: 10.1007/s00134-008-1165-x. Epub 2008 Jun 18. PMID 18563389
- [Background] Murashige D, Jang C, Neinast M, Edwards JJ, Cowan A, Hyman MC, Rabinowitz JD, Frankel DS, Arany Z. Comprehensive quantification of fuel use by the failing and nonfailing human heart. Science. 2020 Oct 16;370(6514):364-368. doi: 10.1126/science.abc8861. PMID 33060364
- [Background] Nielsen R, Moller N, Gormsen LC, Tolbod LP, Hansson NH, Sorensen J, Harms HJ, Frokiaer J, Eiskjaer H, Jespersen NR, Mellemkjaer S, Lassen TR, Pryds K, Botker HE, Wiggers H. Cardiovascular Effects of Treatment With the Ketone Body 3-Hydroxybutyrate in Chronic Heart Failure Patients. Circulation. 2019 Apr 30;139(18):2129-2141. doi: 10.1161/CIRCULATIONAHA.118.036459. PMID 30884964